CLINICAL TRIAL: NCT01048593
Title: A Multicenter, Randomized, Double-masked, Dose-ranging, Phase 2 Study to Evaluate the Efficacy and Safety of IBI-10090 in Cataract Surgery Patients
Brief Title: Efficacy and Safety Study of IBI-10090 in Patients Undergoing Cataract Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated in order to examine study data.
Sponsor: ICON Bioscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C09-01
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Inflammatory Reaction Due to Ocular Lens Prosthesis
Keywords: ocular inflammation cataract surgery; post cataract surgery inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 (Experimental): 114ug
  Interventions: Drug: IBI-10090
- Dose 2 (Experimental): 513ug
  Interventions: Drug: IBI-10090
- Dose 3 (Experimental): 684ug
  Interventions: Drug: IBI-10090

INTERVENTIONS:
Drug: IBI-10090 — Single intraocular injection

SUMMARY:
This study will test the efficacy and safety of IBI-10090 for the reduction of ocular inflammation after cataract surgery.

DETAILED DESCRIPTION:
All patients received active treatment in this study. Dose group 1 received 114ug of dexamethasone, Dose group 2 received 513ug and Dose group 3 received 684ug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 40 years of age scheduled for unilateral cataract surgery (phacoemulsification or extracapsular extraction) with posterior chamber intraocular lens implantation.

Exclusion Criteria:

* Patients who have used any ocular, topical or oral corticosteroids within 7 days prior to Day 0.
* Patients who have used topical ocular NSAIDs in the study eye within 15 days prior to screening.
* Patients with any signs of intraocular inflammation in either eye at screening.
* Patients who have received any prior intravitreal injections in the study eye.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chang, MD, Principal Investigator — Altos Eye Physicians
Locations (1):
- Altos Eye Physicians, Los Altos, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose 1: 114ug dose group
- Dose 2: 513ug dose group
- Dose 3: 684ug dose group
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3
Started | 3 | 2 | 1
Completed | 3 | 2 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Total
Number analyzed (Participants) | 3 | 2 | 1 | 6
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 1 | 6
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — The number of male/female per treatment group was not recorded.
  participants
    Female | 0 | 0 | 0 | 0
    Male | 0 | 0 | 0 | 0
    Unknown | 3 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Anterior Chamber Cells
Description: Efficacy was assessed by slit lamp biomicroscopy to evaluate the anterior chamber cells (ACC) graded on a scale of 0 to 4. The primary efficacy endpoint was complete clearing of ACC, where grade 0 = 0 cells in the anterior chamber on POD 8.
Time Frame: Day 8 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Baseline: Grade 0 (absent) | 3 | 2 | 1
  Baseline: Grade 1 (1-5 cells) | 0 | 0 | 0
  Baseline: Grade 2 (6-15 cells) | 0 | 0 | 0
  Baseline: Grade 3 (16-30 cells) | 0 | 0 | 0
  Baseline: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 8: Grade 0 (absent) | 0 | 0 | 1
  POD 8: Grade 1 (1-5 cells) | 1 | 0 | 0
  POD 8: Grade 2 (6-15 cells) | 1 | 1 | 0
  POD 8: Grade 3 (16-30 cells) | 1 | 1 | 0
  POD 8: Grade 4 (hypopyon) | 0 | 0 | 0

2. Secondary Outcome: Anterior Chamber Flare (ACF) Grade
Description: Efficacy was assessed by slit lamp biomicroscopy to evaluate the anterior chamber flare (ACF) graded on a scale of 0 to 4.
Time Frame: Day 90 post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Baseline: Grade 0 (absent) | 3 | 2 | 1
  Baseline: Grade 1 (trace) | 0 | 0 | 0
  Baseline: Grade 2 (mild intensity) | 0 | 0 | 0
  Baseline: Grade 3 (moderate Intensity) | 0 | 0 | 0
  Baseline: Grade 4 (strong intensity) | 0 | 0 | 0
  POD 1: Grade 0 (absent) | 1 | 1 | 0
  POD 1: Grade 1 (trace) | 0 | 0 | 0
  POD 1: Grade 2 (mild intensity) | 2 | 1 | 1
  POD 1: Grade 3 (moderate Intensity) | 0 | 0 | 0
  POD 1: Grade 4 (strong intensity) | 0 | 0 | 0
  POD 3: Grade 0 (absent) | 1 | 1 | 1
  POD 3: Grade 1 (trace) | 1 | 0 | 0
  POD 3: Grade 2 (mild intensity) | 1 | 1 | 0
  POD 3: Grade 3 (moderate Intensity) | 0 | 0 | 0
  POD 3: Grade 4 (strong intensity) | 0 | 0 | 0
  POD 8: Grade 0 (absent) | 0 | 1 | 1
  POD 8: Grade 1 (trace) | 1 | 0 | 0
  POD 8: Grade 2 (mild intensity) | 1 | 1 | 0
  POD 8: Grade 3 (moderate Intensity) | 1 | 0 | 0
  POD 8: Grade 4 (strong intensity) | 0 | 0 | 0
  POD 15: Grade 0 (absent) | 1 | 1 | 1
  POD 15: Grade 1 (trace) | 1 | 0 | 0
  POD 15: Grade 2 (mild intensity) | 1 | 1 | 0
  POD 15: Grade 3 (moderate Intensity) | 0 | 0 | 0
  POD 15: Grade 4 (strong intensity) | 0 | 0 | 0
  POD 30: Grade 0 (absent) | 3 | 1 | 1
  POD 30: Grade 1 (trace) | 0 | 0 | 0
  POD 30: Grade 2 (mild intensity) | 0 | 1 | 0
  POD 30: Grade 3 (moderate Intensity) | 0 | 0 | 0
  POD 30: Grade 4 (strong intensity) | 0 | 0 | 0
  POD 90: Grade 0 (absent) | 3 | 2 | 1
  POD 90: Grade 1 (trace) | 0 | 0 | 0
  POD 90: Grade 2 (mild intensity) | 0 | 0 | 0
  POD 90: Grade 3 (moderate Intensity) | 0 | 0 | 0
  POD 90: Grade 4 (strong intensity) | 0 | 0 | 0

3. Secondary Outcome: Conjunctival Erythema Grade
Description: Conjunctival erythema was evaluated by slit lamp biomicroscopy graded on a scale of 0 to 3.
Time Frame: Day 90 post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Baseline: Grade 0 (no erythema) | 3 | 2 | 1
  Baseline: Grade 1 (pale reddish bulbar) | 0 | 0 | 0
  Baseline: Grade 2 (red bulbar) | 0 | 0 | 0
  Baseline: Grade 3 (bright red bulbar) | 0 | 0 | 0
  POD 1: Grade 0 (no erythema) | 3 | 1 | 1
  POD 1: Grade 1 (pale reddish bulbar) | 0 | 1 | 0
  POD 1: Grade 2 (red bulbar) | 0 | 0 | 0
  POD 1: Grade 3 (bright red bulbar) | 0 | 0 | 0
  POD 3: Grade 0 (no erythema) | 1 | 2 | 1
  POD 3: Grade 1 (pale reddish bulbar) | 1 | 0 | 0
  POD 3: Grade 2 (red bulbar) | 1 | 0 | 0
  POD 3: Grade 3 (bright red bulbar) | 0 | 0 | 0
  POD 8: Grade 0 (no erythema) | 1 | 2 | 1
  POD 8: Grade 1 (pale reddish bulbar) | 0 | 0 | 0
  POD 8: Grade 2 (red bulbar) | 2 | 0 | 0
  POD 8: Grade 3 (bright red bulbar) | 0 | 0 | 0
  POD 15: Grade 0 (no erythema) | 1 | 1 | 1
  POD 15: Grade 1 (pale reddish bulbar) | 1 | 1 | 0
  POD 15: Grade 2 (red bulbar) | 1 | 0 | 0
  POD 15: Grade 3 (bright red bulbar) | 0 | 0 | 0
  POD 30: Grade 0 (no erythema) | 3 | 2 | 1
  POD 30: Grade 1 (pale reddish bulbar) | 0 | 0 | 0
  POD 30: Grade 2 (red bulbar) | 0 | 0 | 0
  POD 30: Grade 3 (bright red bulbar) | 0 | 0 | 0
  POD 90: Grade 0 (no erythema) | 3 | 2 | 1
  POD 90: Grade 1 (pale reddish bulbar) | 0 | 0 | 0
  POD 90: Grade 2 (red bulbar) | 0 | 0 | 0
  POD 90: Grade 3 (bright red bulbar) | 0 | 0 | 0

4. Secondary Outcome: Corneal Edema Grade
Description: Cornea edema was evaluated by slit lamp biomicroscopy graded on a scale of 0 to 3.
Time Frame: Day 90 post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Baseline: Grade 0 (absent) | 3 | 2 | 1
  Baseline: Grade 1 (mild edema) | 0 | 0 | 0
  Baseline: Grade 2 (moderate edema) | 0 | 0 | 0
  Baseline: Grade 3 (severe edema) | 0 | 0 | 0
  POD 1: Grade 0 (absent) | 3 | 1 | 0
  POD 1: Grade 1 (mild edema) | 0 | 1 | 1
  POD 1: Grade 2 (moderate edema) | 0 | 0 | 0
  POD 1: Grade 3 (severe edema) | 0 | 0 | 0
  POD 3: Grade 0 (absent) | 3 | 1 | 1
  POD 3: Grade 1 (mild edema) | 0 | 1 | 0
  POD 3: Grade 2 (moderate edema) | 0 | 0 | 0
  POD 3: Grade 3 (severe edema) | 0 | 0 | 0
  POD 8: Grade 0 (absent) | 3 | 1 | 1
  POD 8: Grade 1 (mild edema) | 0 | 1 | 0
  POD 8: Grade 2 (moderate edema) | 0 | 0 | 0
  POD 8: Grade 3 (severe edema) | 0 | 0 | 0
  POD 15: Grade 0 (absent) | 3 | 2 | 1
  POD 15: Grade 1 (mild edema) | 0 | 0 | 0
  POD 15: Grade 2 (moderate edema) | 0 | 0 | 0
  POD 15: Grade 3 (severe edema) | 0 | 0 | 0
  POD 30: Grade 0 (absent) | 3 | 2 | 1
  POD 30: Grade 1 (mild edema) | 0 | 0 | 0
  POD 30: Grade 2 (moderate edema) | 0 | 0 | 0
  POD 30: Grade 3 (severe edema) | 0 | 0 | 0
  POD 90: Grade 0 (absent) | 3 | 2 | 1
  POD 90: Grade 1 (mild edema) | 0 | 0 | 0
  POD 90: Grade 2 (moderate edema) | 0 | 0 | 0
  POD 90: Grade 3 (severe edema) | 0 | 0 | 0

5. Secondary Outcome: Anterior Chamber Cell Grade
Description: Anterior chamber cells (ACC) grade was evaluated by slit lamp biomicroscopy graded on a scale of 0 to 4.
Time Frame: Day 90 post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Baseline: Grade 0 (absent) | 3 | 2 | 1
  Baseline: Grade 1 (1-5 cells) | 0 | 0 | 0
  Baseline: Grade 2 (6-15 cells) | 0 | 0 | 0
  Baseline: Grade 3 (16-30 cells) | 0 | 0 | 0
  Baseline: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 1: Grade 0 (absent) | 0 | 0 | 0
  POD 1: Grade 1 (1-5 cells) | 1 | 1 | 0
  POD 1: Grade 2 (6-15 cells) | 2 | 0 | 0
  POD 1: Grade 3 (16-30 cells) | 0 | 1 | 1
  POD 1: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 3: Grade 0 (absent) | 0 | 0 | 0
  POD 3: Grade 1 (1-5 cells) | 0 | 1 | 1
  POD 3: Grade 2 (6-15 cells) | 2 | 0 | 0
  POD 3: Grade 3 (16-30 cells) | 1 | 1 | 0
  POD 3: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 8: Grade 0 (absent) | 0 | 0 | 1
  POD 8: Grade 1 (1-5 cells) | 0 | 1 | 0
  POD 8: Grade 2 (6-15 cells) | 2 | 0 | 0
  POD 8: Grade 3 (16-30 cells) | 1 | 1 | 0
  POD 8: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 15: Grade 0 (absent) | 0 | 0 | 0
  POD 15: Grade 1 (1-5 cells) | 1 | 2 | 1
  POD 15: Grade 2 (6-15 cells) | 2 | 0 | 0
  POD 15: Grade 3 (16-30 cells) | 0 | 0 | 0
  POD 15: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 30: Grade 0 (absent) | 3 | 1 | 1
  POD 30: Grade 1 (1-5 cells) | 0 | 1 | 0
  POD 30: Grade 2 (6-15 cells) | 0 | 0 | 0
  POD 30: Grade 3 (16-30 cells) | 0 | 0 | 0
  POD 30: Grade 4 (hypopyon) | 0 | 0 | 0
  POD 90: Grade 0 (absent) | 3 | 2 | 1
  POD 90: Grade 1 (1-5 cells) | 0 | 0 | 0
  POD 90: Grade 2 (6-15 cells) | 0 | 0 | 0
  POD 90: Grade 3 (16-30 cells) | 0 | 0 | 0
  POD 90: Grade 4 (hypopyon) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dose 1 | Dose 2 | Dose 3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=3) | Dose 2 (N=2) | Dose 3 (N=1)
nasopharyngitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
skin infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
rash (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No